CLINICAL TRIAL: NCT00764387
Title: Contrast-enhanced MRI Examination of Cerebral Neoplastic Enhancing Lesions: Comparison of Diagnostic Efficacy of Gd-DOTA 0.5M and Gadobutrol 1.0 M at 0.1 mmol/kg Body Weight: Intraindividual Comparison Clinical Study.
Brief Title: Contrast Enhanced MRI of the CNS - Patients With Known Cerebral Neoplastic Lesions.
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: 91780; 2007-005693-31 (EudraCT Number); 312021 (Other: Company Internal)
Record Dates: First submitted 2008-07-03; First posted 2008-10-02 (Estimated); Last update posted 2014-12-05 (Estimated); Status verified 2014-12

CONDITIONS: Neoplastic CNS Lesions
Keywords: Neoplastic CNS lesions; Contrast enhanced MRI; Comparison
MeSH Terms: interventions — gadobutrol; gadoterate meglumine

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Arm 1 (Experimental)
  Interventions: Drug: Gadovist® (Gadobutrol, BAY86-4875)
- Arm 2 (Active Comparator)
  Interventions: Drug: Dotarem

INTERVENTIONS:
Drug: Gadovist® (Gadobutrol, BAY86-4875) — 0,1 mmol/kg of body weight in the vein, single administration
  Arms: Arm 1
Drug: Dotarem — 0,1 mmol/kg of body weight in the vein, single administration
  Arms: Arm 2

SUMMARY:
Study to compare of two contrast agents in imaging brain lesions.

ELIGIBILITY:
Inclusion Criteria:

* Known neoplastic CNS lesions

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 166 (Actual)
Dates: Start 2008-03; Primary Completion 2009-05 (Actual); Study Completion 2009-05 (Actual)

PRIMARY OUTCOMES:
The primary analysis will be the comparison of the enhancements characteristics of Gadobutrol and Gd-TOTA on a lesion per lesion basis. | October 2007 to November 2008

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (11):
- Italy (11):
  - Andria, Bari
  - Catania
  - Chieti
  - Messina
  - Milan
  - Napoli
  - Novara
  - Roma
  - Siena
  - Trieste
  - Verona

REFERENCES:
- See also: Click here and search for Bayer Product information provided by EMA — http://www.clinicaltrialsregister.eu